CLINICAL TRIAL: NCT06539936
Title: Regulatory Clearance of the Glide Control Strategy for Upper Limb Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Infinite Biomedical Technologies (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Advanced Arm Dynamics (Unknown)
Responsible Party: Principal Investigator, Rahul Kaliki, Chief Executive Officer, Infinite Biomedical Technologies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R44HD090811 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-08-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Upper Limb
Keywords: amputation; upper limb; myoelectric control; prosthesis; glide

STUDY DESIGN:
Intervention Model Description: Single-Case Experimental Design (SCED)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Multiple Baseline (Experimental): Participants act as their own controls. Participants are fit with a prosthesis system, which includes IBT's Core2 controller, IBT Electrodes, FlexCell batteries, and prosthetic componentry chosen by the patient and their clinical team. The provided controller can operate in two modes of operation: (1) in Direct Control (or DC); and (2) using the Glide control strategy. Participants progress through an AB multiple baseline protocol, where they use the provided prosthesis system for four evaluation periods (totaling 24-weeks in duration). During the A-phase, participants use the system with DC and during the B-phase, participants use the system with the Glide control strategy. For both interventions, the required hardware is the same, while the control software will differ.
  Interventions: Device: Glide; Device: Direct Control

INTERVENTIONS:
Device: Glide — Glide is a myoelectric prosthesis control strategy which enables multifunctional control using a limited set of input EMG signals (as few as two). The Glide control strategy uses the relative contributions of multiple electrode inputs to create a virtual cursor, calculated from a vector summation of multiple EMG channels, to select the type and speed of a movement from a circular map.
Device: Direct Control — Direct Control (DC) is the most common method of control for powered prostheses, which directly links the activity recorded from a single electromyography (EMG) electrode to a prosthesis action. Typically, a pair of EMG electrodes are placed over a pair of agonist/antagonist muscle groups to operate a single DOF (e.g., for transradial amputees the flexor muscles in the forearm may be mapped to the prosthetic hand closing and the forearm extensor muscles mapped to hand opening).

SUMMARY:
The investigators will test the following hypothesis: Use of Glide results in improved functional performance, satisfaction, and usage metrics as compared to use of a standard Direct Control (DC) prosthesis.

This study will compare the use of Glide [Experimental] prosthesis with a DC [Standard] prosthesis in a clinical setting and in unsupervised daily activity. We will follow a multiple baseline design, specifically an AB design. Each of the subjects will use the Experimental and Standard systems over a total of 24-weeks. The A phase is the baseline phase where the DC prosthesis will be used, and the B phase will be the treatment phase where the Glide prosthesis will be used. Participants will undergo an A phase of either 10-weeks, 12-weeks, or 14-weeks duration, with the remaining 14-, 12-, or 10-weeks of the study being dedicated to the B phase.

DETAILED DESCRIPTION:
Recruitment and group assignment: Participants will be recruited through one of Arm Dynamics's six Centers of Excellence. Potentially eligible participants will be identified by their care team and referred to a study team member to go over the details of the patient's involvement and the study protocol. After informed consent and medical clearance are completed, the study prosthetist and occupational therapist will meet with the participant and identify functional goals for their prosthesis. The prosthetist will then begin fabricating the prosthesis. A single prosthesis will be fabricated for use with both control strategies. Switching between control methods will be done through the Glide iPad application. Once fabrication is completed, a clinical team member will configure the assigned control strategy with the subject to achieve maximum functional efficiency.

Prosthesis delivery and occupational therapy (Day 0): After the consenting process and group assignment, patients will return to the clinic to be fit with the prosthesis. Each prosthetic system will include IBT's Glide system, remote electrodes, FlexCell batteries, and prosthetic componentry chosen by the patient and their clinical team. The Glide system also allows for Direct Control of the prosthesis without any hardware change, as long as two of the remote electrodes are positioned according to Direct Control site selection. The fitting process may take multiple visits to adjust the socket. The participant will be given instructions on how to use their prosthesis and activate the various functions of their initial device. Occupational therapy (OT) will be provided over 2 days to the patient to help patients accomplish their desired activities of daily living. At the conclusion of OT, participants will complete baseline assessments of the CAPPFUL, tBBT, CAPROQ, FIT, DASH, and SAM measures.

Phase I DC prosthesis: Over the course of the next 5-, 6-, or 7-weeks, subjects will use their DC prosthesis during their everyday lives. The Glide system is capable of recording usage data during these at-home periods (regardless of which control system is active at a given time). These measures include the Daily Mean Number of Movement Bouts (DMNMB). Using a web portal submission, subjects will report the DMNMB and their Mean Prosthesis Wear Duration (MPWD) for the previous week. At this time, subjects will also complete the CAPROQ and FIT surveys. This data submission will occur weekly.

Phase I Midpoint: Subjects will return to the clinic where they will first complete CAPPFUL, tBBT, CAPROQ, FIT, DASH, and SAM. Once completed, the subject will continue Phase I.

Phase I DC prosthesis: Phase I procedures will be repeated (DC prosthesis).

Crossover checkpoint (Day 70, 84, or 98): Subjects will return to the clinic where they will first complete CAPPFUL, tBBT, CAPROQ, FIT, DASH, and SAM. Once completed, they will have their control strategy transitioned to Glide. They will then receive OT training and complete the same measurements using their prosthesis with Glide control.

Phase II Glide prosthesis: Over the course of the next 7-, 6-, or 5-weeks, subjects will use their Glide prosthesis during their everyday lives. Using the Glide system, subjects will repeat the procedures outlined in Phase I.

Phase II Midpoint: Subjects will return to the clinic where they will first complete CAPPFUL, tBBT, CAPROQ, FIT, DASH, and SAM. Once completed, the subject will continue Phase II.

Phase II Glide prosthesis: Phase II procedures will be repeated (Glide prosthesis).

Endpoint evaluation (Day 168): Measurements from the crossover checkpoint will be made with the Glide prosthesis only. The patient will be re-fit with their pre-study prosthesis, and OT provided as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Trans-radial unilateral limb loss
* Candidate for a multi-articulated myoelectric hand prosthesis as determined by the study prosthetist
* Minimal residual limb length for myoelectric control as determined by the clinical team
* Age of 18 years or greater

Exclusion Criteria:

* Patients with a residual limb that is unhealed from the amputation surgery
* Patients with easily damaged or sensitive skin who would not tolerate EMG electrodes
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Arm Prosthesis and Rehabilitation Outcomes Questionnaire (CAPROQ) | Weekly (i.e., Day 0, Day 7, Day 14, ..., Day 161 and Day 168)
  CAPROQ is a validated patient reported outcome measure that captures key facets of rehabilitation for adults with UL absence or loss: perceived function, satisfaction, and pain. CAPROQ includes a total of 28 questions spread across three sub-scales: 8 satisfaction, 10 perceived functioning, and 10 pain subcategory questions. Responses to all questions are given on a 10-point, Likert-type scale. Higher scores therefore indicate higher levels of overall satisfaction. A singular total CAPROQ score is derived by standardizing each of the CAPROQ subscales and summing these standardized scores together. Higher total scores on the CAPROQ indicate better rehabilitation outcomes and reflect the individual's perceived success with their prosthesis and rehabilitation; specifically, satisfaction with their prosthesis and rehabilitation, greater functional performance, and lesser pain. CAPROQ scores range from 0 to 100.

SECONDARY OUTCOMES:
Capacity Assessment of Prosthesis Performance of the Upper Limb (CAPPFUL) | Baseline (i.e., Day 0); Post-Intervention (i.e., Day 35/42/49, Day 70/84/98, Day 119/126/133, and Day 168)
  CAPPFUL is a validated outcome measure designed as a versatile, low-burden measure of prosthesis performance for any UL functional prosthetic device type and any UL amputation level. CAPPFUL assesses overall performance and 5 functional performance domains during completion of 11 tasks. These require movement in all planes while manipulating everyday objects requiring multiple grasp patterns. Performance domains include control skill, adaptive and maladaptive compensatory movement, component utilization and time for task completion. CAPPFUL scores range from 0 to 100.
Targeted Box and Blocks Tests (tBBT) | Baseline (i.e., Day 0); Post-Intervention (i.e., Day 35/42/49, Day 70/84/98, Day 119/126/133, and Day 168)
  tBBT allows for analysis of movement initiation, grasp, transport, and controlled release of objects. Participant performance in the tBBT is quantified by task completion time. A box with two compartments is used for this assessment. The blocks are arranged in a 4x4 array on the side of the testing hand, using an insert as a guide. Block colors and shapes are correlated to four different grip types available in prosthetic hands. Participants will be instructed to transport one block at a time, starting with the block closest to the partition in the row closest to the participant, placing the blocks in the mirrored position on the opposite side of the partition into target locations defined by an identical insert as on the side of the testing hand. The participant's score will be the time it takes to transport all 16 blocks. Administrators will also keep track of those blocks that are considered unsuccessful transports. tBBT scores start from 0 with no maximum value.
Daily Mean Number of Movement Bouts (DMNMB) | Daily (i.e., Day 0, Day 1, Day 2, ..., Day 167, Day 168)
  DMNMB is an objective measure collected by the controller. The controller does not send any outputs to the prosthesis when the control is in a "rest" state. For all other outputs, movement commands are sent to the prosthesis. Thus, the controller is in a good position to be able to record the amount of prosthesis usage as measured by the frequency of control signals. Such activity is measured in terms of series of continuous movement commands called "movement bouts." The number and length of movement bouts will be recorded and stored in the controller memory. Participants will report DMNMB weekly using a web-based portal.
Mean Prosthesis Wear Duration (MPWD) | Daily (i.e., Day 0, Day 1, Day 2, ..., Day 167, Day 168)
  MPWD measures the mean duration of daily prosthesis wear as a proxy for improved prosthesis acceptance. Prosthesis wear time is defined as the time from when subjects don their prostheses to the time they doff their prostheses and is self-reported by the participant. The log will be provided through a web-based portal and will be filled out weekly, each entry providing the prosthesis wear duration of the previous week.
FIT Survey | Weekly (i.e., Day 0, Day 7, Day 14, ..., Day 161, and Day 168)
  The FIT Survey allows the provider to maximize each patient's comfort, performance, and wear time for uninterrupted use for the life of their prosthesis. After limb loss, the shape and volume of a patient's residual limb will fluctuate throughout their life, potentially impacting comfort, wear time and prosthetic performance. The FIT Survey identifies a patient's residual limb changes in 4 key domains through a low-burden patient reported outcome measure taken every 3 months as a standard of care at Arm Dynamics. Reviewing the Fit Survey weekly during the 24-week research project will allow the clinical team to identify any changes in fit of the prosthesis and immediately address them so that the variables of fit and performance on study results are mitigated.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Baseline (i.e., Day 0); Post-Intervention (i.e., Day 35/42/49, Day 70/84/98, Day 119/126/133, and Day 168)
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a subject-report outcome measure (PROM) developed as a measure of perceived disability in those with upper extremity musculoskeletal disorders. The DASH consists mainly of a 30-item disability/symptom items rated on a 5-point Likert scale, with totals scored 0 (no disability) to 100. It has been validated for the upper limb amputee population.
Speed and Accuracy Measurement | Baseline (i.e., Day 0); Post-Intervention (i.e., Day 35/42/49, Day 70/84/98, Day 119/126/133, and Day 168)
  A Speed and Accuracy Measurement (SAM) will be administered as a simple measurement to identify consistency and accuracy of accessing different components or grasp patterns, as well as speed. This measurement asks the subject to access two predetermined grip patterns OR from access hand then wrist and back 10 times (timed, number of accurate switches out of 10).

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Arm Dynamics, Redondo Beach, California, United States

IPD SHARING:
Plan to Share IPD: No